CLINICAL TRIAL: NCT05930678
Title: Intubation of Obese Patients in the Operating Room With or Without Bag-Mask Ventilation. A Randomized Multicentre Study
Brief Title: Intubation of Obese Patients in the Operating Room With or Without Bag-Mask Ventilation
Acronym: VENT OR NOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC22_0359
Record Dates: First submitted 2023-06-01; First posted 2023-07-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Morbid Obesity; Ventilation Therapy; Complications
MeSH Terms: conditions — Obesity, Morbid | interventions — Masks; Ventilation

STUDY DESIGN:
Intervention Model Description: Morbidly obese patients (BMI greater than or equal to 35).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Without ventilation (Active Comparator): No ventilation sequence during the intubation period and without face mask ventilation during the apnea period
  Interventions: Procedure: No ventilation with face mask
- With ventilation (Experimental): Sequence "with ventilation" during the apnea period with face mask ventilation
  Interventions: Procedure: Ventilation with face mask

INTERVENTIONS:
Procedure: No ventilation with face mask — During the period of apnea (in general anesthesia), the patient did not help with face mask
  Arms: Without ventilation
Procedure: Ventilation with face mask — During the pperiod of apnea (in general anesthesia), the patient did help with face mask
  Arms: With ventilation

SUMMARY:
The aim of the study is to answer a daily question in the operating room: what is the safest technique for intubation of severe/morbid obese patients (BMI 35 or more). There is a great heterogeneity of practices on the subject, so the principle is to determine a common practice to facilitate the management of these patients.

DETAILED DESCRIPTION:
Anesthesia consultation or pre-anesthesia visit:

* screening for inclusion and non-inclusion criteria
* patient information
* collection of consent
* inclusion

D0 (day of inclusion):

* before general anesthesia : collection of epidemiological data (history + clinical examinations) + randomization (Arm A/Not Vent : intubation without ventilation or Arm B/Vent : intubation with ventilation)
* general anesthesia : intubation according to randomization arm + collection primary endpoint + conduct of the intubation procedure + morbidity of the intubation procedure
* after general anesthesia : collection of secondary endpoints + conduct of the intubation procedure + morbidity of the intubation procedure + intraoperative respiratory morbidity
* post-interventional care room : collection of clinical parameters in the ICU : postoperative morbidity + study discharge (hospital discharge)

ELIGIBILITY:
Inclusion criteria:

* patient requiring general anesthesia with intubation for surgery or scheduled endoscopic procedures
* age > 18 years
* with a BMI superior or equal to 35kg.m-²
* patient having signed an informed consent

Non-inclusion criteria:

* ambient air saturation <90%
* urgent surgery < 24 hours
* cardio-thoracic surgery
* mask ventilation not possible (e.g. ATCD, cervical irradiation, fixed mandible)
* formal contraindication to mask ventilation (e.g. occlusive syndrome, non fasting patient, symptomatic gastroesophageal reflux untreated or persistent under treatment)
* wish of the operator for high flow oxygen preoxygenation
* wish of an intubation without curare by the operator
* pregnant or breast-feeding women
* protected adults (guardianship, curatorship or safeguard of justice)
* participation in another randomized clinical research study concerning preoxygenation and relevant to the primary endpoint
* absence of affiliation to the French social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of an intubation sequence "with ventilation during apnea" versus a sequence "without ventilation during apnea" in preventing complications related to intubation of the obese patient in the operating room | From induction of general anesthesia to 10 minutes after intubation
  Comparison of the incidence of intubation-related complications. Complications identified for the primary endpoint will be: desaturations < 95%, need for 2 or more intubation attempts (including alternative technique), occurrence of inhalation/regurgitation or hypotension with systolic blood pressure < 80 mmHg, with or without amine. Complications will be recorded from induction of general anesthesia to 10 minutes after intubation

SECONDARY OUTCOMES:
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 8 hours
  Difficulty with mask ventilation (yes/no)
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 10 minutes
  Measure of the saturation before the first laryngoscopy with oximeter
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 10 minutes
  Measure of the lowest saturation during the intubation procedure and the following 10 minutes
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 8 hours
  Quality of exposure under laryngoscopy (position of the patient)
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 8 hours
  Difficulties in intubation (yes/no)
Impact of the nature of the intubation sequence on the progress of the intubation procedure between patient with face mask and patient without face mask | During the general anesthesia, up to 8 hours
  Description of intubation (mandrin, videolaryngoscope, videolaryngoscope)
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Rate of desaturation <80% (yes/no)
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Rate of desaturation <90% (yes/no)
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Presence of severe hypotension during intubation and in the following hour defined by a systolic blood pressure < 80 mmHg, with or without amine (yes/no)
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Number of participants with cardiac arrest
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Death during intubation
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Difficulties in intubations (yes/no) with the number of intubation attempts
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Number of participants with cardiac rhythm disorders
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Number of participants with esophageal intubations
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Number of participants with regurgitation/inhalation
Impact of the nature of the intubation sequence on morbidity related to the intubation procedure between patient with face mask and patient without face mask | up to 8 hours
  Number of participants with dental breaks
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | 5 minutes, 30 minutes and 1 hour after intubation
  Need for FiO2 >50% during surgery to achieve >95% saturation (yes/no)
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Length of stay in the post-operation monitoring room
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Duration of postoperative mechanical ventilation(in minutes)
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Number of participants with nausea
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Number of participants with vomiting
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Length of hospitalization since randomization
Impact of the nature of the intubation sequence on immediate intraoperative and postoperative respiratory morbidity between patient with face mask and patient without face mask | up to 28 days
  Hospital discharge status (dead/alive)

CONTACTS AND LOCATIONS:
Overall Officials: Mickael VOURC'H, PhD, Principal Investigator — Nantes University Hospital
Locations (13):
- France (13):
  - CHU Nantes, Nantes, Loire Atlantique
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - CHU de Dijon, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - HCL - Hôpital Edouard Herriot, Lyon
  - CHU de Nantes - site Laennec, Nantes
  - CHU de Rennes, Rennes
  - CH de Saint-Nazaire, Saint-Nazaire
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU Toulouse, Toulouse
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Znaidi S, Deransy R, Asehnoune K, Le Penndu M, Rozec B, Jumel G, Lasocki S, Cadic-Pelletier A, Guinot PG, Duchalais A, Cirenei C, Abrard S, Beloeil H, Fortuit C, Landrin J, Porta Bonete G, Defrancq F, Pere M, Vourc'h M. Intubation of obese patients in the operating room with or without bag-mask ventilation: study protocol for a randomized multicenter trial (VENT OR NOT). Trials. 2025 Nov 11;26(1):492. doi: 10.1186/s13063-025-09114-z. PMID 41219812